CLINICAL TRIAL: NCT01078467
Title: The Molecular Anatomy of Oral Wound Healing
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100020; 10-D-0020
Record Dates: First submitted 2010-02-27; First posted 2010-03-02 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-02-19

CONDITIONS: Wounds and Injuries; Wound Healing; Ulcer
Keywords: Wound Healing; Oral Wounds; Cutaneous Wounds; Gene Array Analysis; Proteomic Analysis; Healthy Volunteer; HV
MeSH Terms: conditions — Wounds and Injuries; Ulcer

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Two important properties distinguish the healing process of skin wounds from that of wounds of the mucous membranes of the mouth (oral mucosa). Although the skin and the oral mucosa tissues are similar in nature, oral mucosa have more rapid healing and a lack of scar tissue formation. However, oral wound healing in general has been poorly studied, and more information is needed to determine how specific aspects of the oral environment affect the healing process.
* Researchers are interested in identifying various factors that contribute to oral wound healing. Studying this process would help researchers explore procedures to accelerate the healing of critically-sized oral lesions formed by trauma, surgery, radiation therapy, infection, and other damage to the mouth. In addition, research into scar-free healing could be applied to other mucosal sites to promote healing and minimize unsightly scars that may compromise the tissue.

Objectives:

- To identify the specific factors that enable rapid and nearly scar-free healing of oral mucosa.

Eligibility:

* Healthy male volunteers between 18 and 40 years of age.
* Regular cigarette, cigar, and pipe smokers; occasional smokers who smoke more than 1 day a week or have smoked in the prior month; users of chewing tobacco or betel nut; and heavy drinkers (three or more alcoholic drinks per day) will be excluded.

Design:

* Participants will have a medical history and examination, and will provide blood samples at the start of the study.
* Participants will provide oral mucosa samples from the inside of the cheek, taken using a dermal punch. At the same time, participants will provide skin biopsy samples of approximately the same size. After the skin and oral mucosa samples are taken, participants will be divided into three groups for follow-up procedures.
* Group 1: No further samples will be collected. This group will help document the normal healing process.
* Group 2: A second, slightly larger biopsy, which will include the area of the first biopsy, will be taken on day 3. Both skin and oral mucosa biopsies will be taken.
* Group 3: A second, slightly larger biopsy will be taken on day 6, in a similar way as described for Group 2. Both skin and oral mucosa biopsies will be taken.
* Wounds will be photographed with a digital camera on days 3, 6, 9, 13, and 15; and the healing will be monitored at the scheduled clinic visits.

DETAILED DESCRIPTION:
BACKGROUND:

Two important properties distinguish the process of healing of oral mucosa wounds from those of the skin: more rapid healing and the absence of scar tissue formation. This is remarkable given the apparent similarities of the two tissues. There are, however, prominent differences in the healing environment, such as hydration, growth factor availability, inflammatory response, and microbial exposure. Knowledge as to the causal contribution of each of these factors to the differential healing response of the two epithelia is mostly anecdotal, and oral wound healing has generally been poorly studied. This study seeks to provide a global molecular definition of oral wound healing in comparison to that of the skin. The overall aim will be to identify the specific factors that enable rapid and nearly scar-free healing of oral mucosa. Identification of these physiological and molecular determinants will have widespread implications for human oral health. Among others, it would provide venues for the targeted exploration of procedures to accelerate the healing of critically-sized oral lesions formed by trauma, surgery, radiation therapy, infection, and other oral pathologies, which, if untreated, lead to permanent disability and dysfunction. Moreover, pathways and/or molecules identified in these studies which may facilitate rapid, scar-less healing could be considered for application to non-oral mucosal sites to promote healing and minimize unsightly scars, which may also compromise the functional integrity of the tissue.

Hypotheses:

* There are significant differences in gene and protein expression between wound healing in skin and oral mucosa.
* The recruitment of inflammatory cells associated with a large up-regulation of inflammation-associated genes, including cytokines and chemokines, in the epithelial cells of skin wounds may account for these differences.
* There are specific gene programs that can explain the presence of significant scarring in skin tissues but not in oral mucosa.

OBJECTIVES:

The overall objective of this pilot study proposal is to establish the gene and protein expression profiles during the early stages (1-6 days) of normal oral wound repair. By comparing these profiles with those of cutaneous wound healing, we may be able to identify molecules exclusive to oral wound repair that could represent biomarkers of the healing process or serve as new therapeutic targets in pathological wound healing and cancer. One specific hypothesis to be tested is that the level of expression of pro-inflammatory gene networks by wound-infiltrating keratinocytes constitutes the most significant difference between the human oral and cutaneous wound transcriptomes. The specific hypothesis has been developed from data obtained from our recent complementary oral and skin wound healing studies in animals.

ELIGIBILITY:

Healthy male volunteers age 18 to 40 will be enrolled in this study.

DESIGN:

Oral mucosa samples: A sterile 3-mm dermal punch will be used to create uniform, full-thickness biopsy in the mucosa of the cheek just above the occlusal plane. Circular pieces of tissue of approximately 2 mm in depth will be removed on the day of biopsy (day 1). These subjects will be subsequently be randomly grouped as follows:

Group 1: no further samples will be collected; pictures will be taken on days 3, 6, 9, 13, and 15 (see Timetable). This group will help document the normal healing process under the conditions of the present study, including the lack of scaring in the area selected for the initial wound in the oral mucosa as compared with the skin.

Group 2: a second biopsy will be taken on day 3, which will include the area of the first biopsy with sterile 5 mm punch, following the same procedure as described for day 0; pictures will be taken according to the schedule set in the Timetable. This second biopsy will enabled sampling the healing area induced by the first biopsy. By selecting a punch size two millimeters wider and taking a sample concentric to the first one, we can assure complete removal of the area of interest.

Group 3: a second biopsy will be taken on day 6, respectively, in a similar way as described for Group 2; pictures will be taken according to the Timetable.

Skin samples: In parallel to the oral biopsies, skin biopsies of similar size and depth as the oral biopsy from the same subjects will be obtained from the axillary region following the same schedule and procedure, including a second biopsy for groups 2 and 3.

Wounds will be photographed with a digital camera and the healing monitored at clinic visits per schedule above. The excised tissues in each case will be immediately bisected on ice; half of the sample will be fixed in 4% formaldehyde/PBS and embedded in paraffin for standard histology and immunohistochemistry, and the remaining half will be placed in OCT-filled plastic base molds, flash frozen in liquid nitrogen, and stored at 80 (Infinite)C until processed for genomic and proteomic analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy male volunteers age 18 to 40.
* All volunteers must sign informed consent indicating their understanding that specimens and demographic information will be collected solely for research purposes.

EXCLUSION CRITERIA:

Subjects with known inflammatory, chronic, and infectious diseases. These conditions include but are not limited to:

* Diabetes
* Heart failure
* Pulmonary disease
* Rheumatoid arthritis
* Systemic lupus erythematosus
* Sarcoidosis
* Sj(SqrRoot)(Delta)grens syndrome
* Dermatomyositis
* Psoriasis
* Cellulitis

Patients with known bleeding disorders or conditions associated with bleeding. These conditions include but are not limited to:

* Hemophilia
* von Willebrand disease
* Protein C/S deficiency
* Antithrombin III deficiency
* Liver disease
* Patients on medications that interfere with blood clotting or blood thinners. These medications include but are not limited to: ibuprofen aspirin, warfarin (Coumadin), ticlopidine (Ticlid), clopidogrel (Plavix), and others.
* Subjects with clinically significant abnormal laboratory values will be ineligible

Complete blood count (CBC)

Platelet level: <100 - >500/ 10(3)/mcL<TAB>

Hemoglobin: <10; > 17.5gr/L<TAB>

Hematocrit: <30; >51%<TAB>

White blood cell count: <3; >12 10(3)/mcL

Partial thromboplastin time: <20; >42 sec

Prothrombin time: <10; >20 sec

C-reactive protein: > 4 mg/L

Erythrocyte sedimentation rate: >40 ml/h

* Recent unintentional weight loss of >10 lbs over the past 6 weeks prior to screening
* Have undergone general or oral surgery within the last 30 days
* Treated with systemic steroids in the past 12 months
* Subjects with a history of abnormal scar formation (i.e., keloids, hypertrophic scarring)
* Subjects who have used tobacco products and/or betel nut within one month of the screening evaluation. Tobacco products include cigarette, pipe, cigar, and chewing tobacco
* Heavy drinkers defined as drinking greater than or equal to alcoholic drinks per day
* Subjects that, at the oral clinical examination, show any of the nonmalignant lesions associated with heavy smoking/tobacco chewing will be excluded. These findings include but are not limited to:
* Tooth stains
* abrasions
* smoker s melanosis
* acute necrotizing gingivitis
* burns
* erythematous or keratotic patches
* black hairy tongue
* nicotinic stomatitis
* palatal erosions
* Subjects with preneoplastic (leukoplakia, erythroplakia, submucous fibrosis) or neoplastic lesions
* Subjects with known or suspected allergies or adverse reactions to any of the agents used for skin preparation, local anesthesia, or pain control or with known or suspected allergy or adverse reaction to Prolene (polypropylene) sutures

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2010-02-02; Study Completion 2019-02-19

CONTACTS AND LOCATIONS:
Overall Officials: Janice S Lee, DDS, MD, Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schafer M, Werner S. Transcriptional control of wound repair. Annu Rev Cell Dev Biol. 2007;23:69-92. doi: 10.1146/annurev.cellbio.23.090506.123609. PMID 17474876
- [Background] Baker H, Patel V, Molinolo AA, Shillitoe EJ, Ensley JF, Yoo GH, Meneses-Garcia A, Myers JN, El-Naggar AK, Gutkind JS, Hancock WS. Proteome-wide analysis of head and neck squamous cell carcinomas using laser-capture microdissection and tandem mass spectrometry. Oral Oncol. 2005 Feb;41(2):183-99. doi: 10.1016/j.oraloncology.2004.08.009. PMID 15695121
- [Background] Lee HG, Eun HC. Differences between fibroblasts cultured from oral mucosa and normal skin: implication to wound healing. J Dermatol Sci. 1999 Nov;21(3):176-82. doi: 10.1016/s0923-1811(99)00037-7. PMID 10527379